CLINICAL TRIAL: NCT01588522
Title: Phase I Dose-Escalation Study, to Evaluate the Safety, Tolerability and Pharmacokinetics of a Topical Compound 31543 (Calcitriol, USP) in Adult Cancer Patients Receiving Taxane-based Chemotherapy Regimens for the Treatment of Advanced or Recurrent Disease
Brief Title: Compound 31543 (Calcitriol, USP) in Patients Receiving Taxane-based Chemotherapy Regimens for the Treatment of Chemotherapy-Induced Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CTL0211
Record Dates: First submitted 2012-04-20; First posted 2012-05-01 (Estimated); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy-Induced Alopecia
Keywords: alopecia
MeSH Terms: conditions — Alopecia | interventions — Calcitriol

STUDY DESIGN:
Intervention Model Description: A standard 3+3 dose escalation design was employed, over 6 dose levels, with 3 to 6 patients at each dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Compound 31543 Calcitriol - 5 μg/mL (Experimental): Compound 31543 Calcitriol (5 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 5 μg/mL
- Compound 31543 Calcitriol - 10 μg/mL (Experimental): Compound 31543 Calcitriol (10 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 10 μg/mL
- Compound 31543 Calcitriol - 20 μg/mL (Experimental): Compound 31543 Calcitriol (20 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 20 μg/mL
- Compound 31543 Calcitriol - 40 μg/mL (Experimental): Compound 31543 Calcitriol (40 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 40 μg/mL
- Compound 31543 Calcitriol - 60 μg/mL (Experimental): Compound 31543 Calcitriol (60 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 60 ug/mL
- Compound 31543 Calcitriol - 80 μg/mL (Experimental): Compound 31543 Calcitriol (80 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
  Interventions: Drug: Compound 31543 Calcitriol 80 μg/mL

INTERVENTIONS:
Drug: Compound 31543 Calcitriol 5 μg/mL — 5 μg/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 5 μg/mL
Drug: Compound 31543 Calcitriol 10 μg/mL — 10 μg/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 10 μg/mL
Drug: Compound 31543 Calcitriol 20 μg/mL — 20 μg/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 20 μg/mL
Drug: Compound 31543 Calcitriol 40 μg/mL — 40 μg/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 40 μg/mL
Drug: Compound 31543 Calcitriol 60 ug/mL — 60 ug/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 60 μg/mL
Drug: Compound 31543 Calcitriol 80 μg/mL — 80 μg/mL Topical Solution
  Other Names: Calcitriol; BPM31543 Topical Solution
  Arms: Compound 31543 Calcitriol - 80 μg/mL

SUMMARY:
The goal of this clinical trial is to learn if Compound 31543 (topical calcitriol) for treatment of hair-loss in patients with a diagnosis of breast cancer, gynecologic cancer or sarcomas receiving a taxane-based chemotherapy is safe. The main questions it aims to answer are:

* What medical problems do participants have when using compound 31543?
* How much Compound 31543 is in blood after treatment?
* How much hair is lost during treatment?

Participants will:

* Apply Compound 31543 to their scalp twice a day, starting at least 5 days before starting chemotherapy for at least 3 months or until chemotherapy treatment is completed.
* Have blood drawn on weeks 1, 5, 9, 13, and 54.
* Have photographs taken of their hair before starting and at weeks 7, 15, 27, and 54.
* Keep a diary of the condition of their hair.

DETAILED DESCRIPTION:
This was a multi-center, single arm, dose-escalation Phase 1 study to determine the maximum tolerated dose (MTD), PK, and the overall safety and tolerability of Compound 31543 in patients with a diagnosis of early-stage or locally advanced, unresectable and/or metastatic cancer, or patients with operable cancer, who were scheduled to receive follow up treatment with a taxane-based chemotherapy regimen, as per the physician's discretion. A standard 3+3 dose escalation design was employed, over 6 dose levels, with 3 to 6 patients at each dose level. Eligible patients in each cohort, >18 years of age and scheduled to receive a taxane-based regimen with treatment breaks as per physician's discretion, initially received or applied the topical formulation of Compound 31543 to the scalp twice daily either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).To determine the MTD for Compound 31543, dose escalation was conducted in stepwise increments, in the absence of dose-limiting toxicity (DLT) defined as clinically significant Grade 3 or 4 non-hematologic toxicity assessed as possibly, probably, or definitely related to Compound 31543 and not to the taxane-based chemotherapy, as best determined by investigator; assessment of DLTs was made weekly during the first 28 days of Compound 31543 treatment and subsequently thereafter every 4 weeks.

Pharmacokinetic (PK) data were evaluated for each dose level before escalation of Compound 31543 to the next dose level in all patients. PK blood samples were collected on Day 1 prior (pre-dose) to the first-morning dose of topical Compound 31543 and at 2, 4, and 8 hours post-dose after the first application of Compound 31543 on Day 1. PK samples were also collected 12 hours after the last, evening dose of Compound 31543 (i.e., before the first Day 1 of the next 28-day treatment) on Weeks 5, 9, 13, and 54.

Potential efficacy of the Compound 31543 was evaluated by photographic assessments and self-assessment diaries performed at baseline and Weeks 7, 15, 27, and 54. Photographic assessments were performed using a Canon digital camera system on views of the front of head/face, bilateral sides of head, and back and top of head/scalp view, as well as close-up photographs of a superior view and a vertex view with hair parted in the center and combed away from the part. Photographs were standardized for lighting, camera angle, and position to the participant's head.

Additionally, patients maintained a medication application diary and a self-assessment diary. The patient completed diary collected patient-reported assessments of hair thickness, fullness, volume, breakage, and cosmetic qualities (ease of styling, etc.) based on a 10-point analog scale for each parameter/question during the first 15 weeks after initiating calcitriol Compound 31543 and at Weeks 19, 23, and 27.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* Able to fully understand and participate in the informed consent process
* Patients who are scheduled to receive a taxane-based regimen for a histologically confirmed solid tumor that is:

  1. Early stage and/or treatment naïve, or
  2. Relapsed or is refractory to previous therapy, or
  3. Operable and necessitates adjuvant or neo-adjuvant treatment
* Have no evidence of alopecia or mild alopecia (NCI CTCAE v.4.0 grade 1 alopecia defined as hair loss of <50% of normal for that individual that is not obvious from a distance but only on close inspection; a different hair style may be required to cover the hair loss but it does not require a wig or hair piece to camouflage). Female/male-pattern baldness or age-related hair loss are allowed if not greater than grade 1, per NCI-CTCAE v. 4.0. Patients that have previously lost their hair may enroll if they currently have Grade 0 or 1 alopecia
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1 within 14 days prior to registration
* Has baseline neutrophil counts of > 1500 cells/mm3 within 72 hours prior to registration
* Has serum calcium less than or equal to upper limit of normal (ULN) (for patients with an albumin lower than 3.0, a corrected calcium serum calcium = serum calcium +[0.8][3.5-serum albumin]) within 72 hours prior to registration

Exclusion Criteria:

* Patients receiving calcium-lowering therapy or drugs that may affect calcium levels (e.g., calcitonin, mithramycin, phosphate, denosumab) within 4 weeks of initiation of topical calcitriol. Patients who have been managed with bisphosphonates or calcium-lowering therapy for 3 months or greater prior to the start of the trial and have demonstrated evidence for stability of calcium metabolism would be considered eligible for participation in the trial.
* Has a history of drug or alcohol abuse within 1 year of study enrollment as determined by the investigator.
* Patients who elect to shave the scalp hair prior to the initiation of chemotherapy or who plan to do so during the chemotherapy treatment.
* Any dermatological condition that in the opinion of the investigator will affect the absorption of the study medication, e.g. Atopic Dermatitis, etc.
* Has been treated with an investigational agent within 30 days or six half-lives of its biologic activity whichever is longer, before the start of study. (Patients may not be concurrently enrolled on another trial or concurrently treated with another investigational agent)
* Patients with a history of hypercalcemia or vitamin D toxicity, or hospitalization for treatment of angina, myocardial infarction, or congestive heart failure or psychiatric illness currently or within 30 days of study entry as determined by the investigator.
* Has a history of significant allergy to calcitriol as determined by the investigator.
* Has any condition that interferes with the ability of the subject to understand or comply with the requirements of the study.
* Patients taking Vitamin D supplements during the study, unless they have been taking Vitamin D supplements for 30 days or more prior to the start of the study and that the dose of the Vitamin D supplement remain the same throughout the study.
* Patients treated with medications that are known to affect calcium levels within 4 weeks of initiation of topical therapy (>500 IU vitamin A, calcium supplements, fluoride, antiepileptics).with the exception of patients on stable therapy for more than six months
* Patients with hypercalcemia or kidney stones
* Patients that indicate they have significant hair breakage or hair damage and associated hair loss from hair over-processing within the last 30 days due to peroxide applications, permanent hair coloring, bleaches, streaking, perms, relaxers and/or hair oxidative dyes.
* Current alopecia grade 2 or greater as per NCI-CTCAE v.4.0, or significant hair loss or hair breakage
* Prior radiation to the cranium
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Lacouture, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Monica Mita, MD, Principal Investigator — Samuel Oschin Comprehensive Cancer Institute Cedars-Sinai
Locations (2):
- United States (2):
  - Samuel Oschin Comprehensive Cancer Institute Cedars-Sinai, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 2 US sites
Pre-assignment Details: Patients scheduled to receive follow up treatment with a taxane-based chemotherapy regimen
Groups:
- Compound 31543 Calcitriol - 40 μg/mL: Compound 31543 Calcitriol (40 μg/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
Period: Overall Study
Arm/Group | Compound 31543 Calcitriol - 5 μg/mL | Compound 31543 Calcitriol - 10 μg/mL | Compound 31543 Calcitriol - 20 μg/mL | Compound 31543 Calcitriol - 40 μg/mL | Compound 31543 Calcitriol - 60 μg/mL | Compound 31543 Calcitriol - 80 μg/mL
Started (All patients enrolled (signed the informed consent form).) | 3 | 5 | 6 | 5 | 6 | 3
Treated (All patients who received at least one application of Compound 31543 Calcitriol.) | 3 | 3 | 6 | 4 | 4 | 3
Completed (All patients that completed three 28 day cycles of Compound 31543 Calcitriol.) | 1 | 0 | 2 | 2 | 2 | 3
Not Completed | 2 | 5 | 4 | 3 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 3 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Grade 2 alopecia | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Severe toxicity of chemotherapy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Taken off taxane-based regimen | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did not initiate chemotherapy | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Received at least 1 dose of Compound 31543 Calcitriol
Groups:
- Compound 31543 Calcitriol - 5 ug/mL: Compound 31543 Calcitriol (5 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Compound 31543 Calcitriol - 10 ug/mL: Compound 31543 Calcitriol (10 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Compound 31543 Calcitriol - 20 ug/mL: Compound 31543 Calcitriol (20 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Compound 31543 Calcitriol - 40 ug/mL: Compound 31543 Calcitriol (40 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Compound 31543 Calcitriol - 60 ug/mL: Compound 31543 Calcitriol (60 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Compound 31543 Calcitriol - 80 ug/mL: Compound 31543 Calcitriol (80 ug/mL), Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications either for 2 weeks or 7 ± 2 days (if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily for the duration of the individual patient's chemotherapy (up to a maximum of 54 weeks).
- Total: Total of all reporting groups
Arm/Group | Compound 31543 Calcitriol - 5 ug/mL | Compound 31543 Calcitriol - 10 ug/mL | Compound 31543 Calcitriol - 20 ug/mL | Compound 31543 Calcitriol - 40 ug/mL | Compound 31543 Calcitriol - 60 ug/mL | Compound 31543 Calcitriol - 80 ug/mL | Total
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 4 | 3 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (8.5) | 47.0 (6.08) | 54.0 (12.98) | 51.0 (17.83) | 47.3 (18.46) | 58.0 (12.17) | 51.7 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 4 | 4 | 3 | 23
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 2 | 3 | 6 | 3 | 3 | 2 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 2
  White | 3 | 2 | 5 | 3 | 3 | 3 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLT) of Topical Compound 31543
Description: DLTs were graded according to the CTCAE v4.0. A DLT was defined as a clinically significant Grade 3 or 4 (severe or life-threatening, respectively) non-hematologic toxicity occurring during the first 28-day treatment cycle, and determined to be possibly, probably, or definitely related to BPM31543 and not the taxane-based regimen as best determined by investigators.
Time Frame: 28 days
Population: Consisted of all patients who received at least one application of Compound 31543.
Measure: Count of Participants; unit: Participants
Groups:
- Compound 31543 Calcitriol - 5 μg/mL; Compound 31543 Calcitriol - 10 μg/mL; Compound 31543 Calcitriol - 20 μg/mL; Compound 31543 Calcitriol - 40 μg/mL; Compound 31543 Calcitriol - 60 μg/mL; Compound 31543 Calcitriol - 80 μg/mL: Compound 31543 Calcitriol, Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications
Arm/Group | Compound 31543 Calcitriol - 5 μg/mL | Compound 31543 Calcitriol - 10 μg/mL | Compound 31543 Calcitriol - 20 μg/mL | Compound 31543 Calcitriol - 40 μg/mL | Compound 31543 Calcitriol - 60 μg/mL | Compound 31543 Calcitriol - 80 μg/mL
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pre-dose Concentrations of Compound 31543
Description: Pre-dose concentrations of Compound 31543 from serum samples collected on Week 1 Day 1.
Time Frame: pre-dose on day 1 of Week 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Compound 31543 Calcitriol - 5 ug/mL | Compound 31543 Calcitriol - 10 ug/mL | Compound 31543 Calcitriol - 20 ug/mL | Compound 31543 Calcitriol - 40 ug/mL | Compound 31543 Calcitriol - 60 ug/mL | Compound 31543 Calcitriol - 80 ug/mL
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 2 | 3
pg/mL | 49.0 (5.8) | 43.2 (14.8) | 54.3 (31.5) | 58.4 (19.4) | 32.8 (5.2) | 37.8 (15.5)

3. Secondary Outcome: Cmax of Compound 31543 on Week 1 Day 1
Description: Cmax of Compound 31543 was calculated using serum samples collected on Week 1 Day 1 pre-dose and at 2 ± 0.5 hours, 4 ± 0.5 hours, and 8 ± 1 hours post-dose. The 8-hour Week 1 Day 1 sample was collected before the second of the daily doses.
Time Frame: 8 hours
Population: Pharmacokinetic Parameters for Serum Calcitriol Concentrations on Week 1, Day 1 of BPM31543 Administration (PK Population)
  The pharmacokinetic evaluable population was intended to include all patients with concentration results for the four samples scheduled for Week 1 Day 1.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- 5 μg/mL; 10 μg/mL; 20 μg/mL; 40 μg/mL; 60 μg/mL; 80 μg/mL: BPM1543 Calcitriol, Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 2 | 2
pg/mL | 51.6 (6.9) | 47.2 (13.6) | 42.5 (8.5) | 81.0 (8.1) | 36.0 (9.8) | 53.5 (16.1)

4. Secondary Outcome: AUC0-t of Compound 31543 on Week 1 Day 1
Description: Area under the curve (AUC0-t) of Compound 31543 was calculated from serum samples collected on Week 1 Day 1 pre-dose and at 2 ± 0.5 hours, 4 ± 0.5 hours, and 8 ± 1 hours post-dose. The 8-hour Week 1 Day 1 sample was collected before the second of the daily doses.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: pg•hour/mL
Arm/Group | Compound 31543 Calcitriol - 5 ug/mL | Compound 31543 Calcitriol - 10 ug/mL | Compound 31543 Calcitriol - 20 ug/mL | Compound 31543 Calcitriol - 40 ug/mL | Compound 31543 Calcitriol - 60 ug/mL | Compound 31543 Calcitriol - 80 ug/mL
Number analyzed (Participants) | 3 | 2 | 3 | 2 | 2 | 2
pg•hour/mL | 346 (10) | 334 (163) | 259 (60) | 530 (165) | 230 (87) | 370 (99)

5. Secondary Outcome: Top View Photographic Review Score
Description: Top of head/scalp view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: Evaluable Population defined as all patients who completed at least one photographic assessment and diary completion through Week 7. Some patients discontinued treatment prior to week 15 and are therefore only analyzed at week 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 2 | 3
score on a scale
  Week 7 | -1 (0) | -1.5 (0.71) | -1 | -3 (0) | -1 (0) | -2 (1)
  Week 15: number analyzed (Participants) | 1 | 0 | 1 | 1 | 2 | 2
  Week 15 | -2 |  | -1 | -3 | -2 (1.41) | -3 (0)

6. Secondary Outcome: Right Side Photographic Review Score
Description: Right side of head/scalp view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 2 | 3
score on a scale
  Week 7 | -1 (0) | -2 | -1 (0) | -2.3 (1.15) | -1 (0) | -1.7 (0.58)
  Week 15: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 3
  Week 15 | -2 |  | -1.5 (0.71) | -3 | -2 (1.41) | -2.5 (.71)

7. Secondary Outcome: Left Side Photographic Review Score
Description: Left side of head/scalp view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 3
score on a scale
  Week 7 | -0.5 (0.71) | -1 (0) | -1 (0) | -2.3 (1.15) | -1 (0) | -1.7 (0.58)
  Week 15: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 2
  Week 15 | -2 |  | -1.5 (0.71) | -3 | -2 (1.41) | -2.5 (0.71)

8. Secondary Outcome: Front Photographic Review Score
Description: Front of head/face view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 3
score on a scale
  Week 7 | -0.5 (0.71) | -0.5 (0.71) | -1 (0) | -1.7 (0.58) | -1 (0) | -2.3 (0.58)
  Week 15: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 2
  Week 15 | -2 |  | -1.5 (0.71) | -2 | -2 (1.41) | -2.5 (0.71)

9. Secondary Outcome: Back Photographic Review Score
Description: Back of head/face view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 3
score on a scale
  Week 7 | -0.5 (0.71) | -0.5 (0.71) | -1 (0) | -2 (1) | -1 (0) | -2 (1)
  Week 15: number analyzed (Participants) | 1 | 0 | 2 | 1 | 2 | 2
  Week 15 | -2 |  | -1 (0) | -3 | -2 (1.41) | -2.5 (0.71)

10. Secondary Outcome: Superior (Mid Pattern) Photographic Review Score
Description: Mid-pattern of the scalp from a superior view at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 2 | 3
score on a scale
  Week 7 | -1 | -1 (0) | -1 (0) | -1.7 (0.58) | -0.5 (0.71) | -1.7 (0.58)
  Week 15: number analyzed (Participants) | 0 | 0 | 2 | 1 | 2 | 2
  Week 15 |  |  | -1 (0) | -2 | -2 (1.41) | -2.5 (0.71)

11. Secondary Outcome: Vertex Photographic Review Score
Description: Vertex view with hair parted in the center at 7 and 15 weeks were compared to baseline images and scored on a 7-point evaluation scale: -3 = >75% great hair loss; -2 = 50-75% moderate hair loss; -1 = 25-49% slight hair loss; 0 = 0-24% hair loss/gain, 1 = 25-49% slight hair gain; 2 = 50-75% moderate hair gain; 3 = >75% greatly increased/hair gain.
Time Frame: 7 and 15 weeks
Population: Evaluable Population defined as all patients who completed at least one photographic assessment and diary completion through Week 7. Not all patients had this photograph taken. Some patients discontinued treatment prior to week 15 and are therefore only analyzed at week 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 μg/mL | 10 μg/mL | 20 μg/mL | 40 μg/mL | 60 μg/mL | 80 μg/mL
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 2 | 3
score on a scale
  Week 7 |  |  | -1 (0) | -1.7 (0.58) | -0.5 (0.71) | -1.7 (0.58)
  Week 15: number analyzed (Participants) | 0 | 0 | 2 | 1 | 2 | 2
  Week 15 |  |  | -1 (0) | -2 | -1.5 (2.12) | -2.5 (0.71)

ADVERSE EVENTS:
Time Frame: 2 weeks (or 7 days ± 2 days if the patient was unable or unwilling to undergo 2 weeks of pre-treatment) prior to the first dose of chemotherapy and continued the application twice daily until termination of chemotherapy treatment (up to a maximum of 54 weeks)
Description: Safety assessments included treatment-emergent adverse events (TEAEs) and change from baseline (CFB) for vital signs (blood pressure, temperature, respiration rate, heart rate), physical examinations including weight, and laboratory tests (NCI-CTCAE v4.0) at Weeks 1, 2, 3, 5, 7, 11, 15, 27, and 54.
Groups:
- Compound 31543 Calcitriol - 5 μg/mL; Compound 31543 Calcitriol - 10 μg/mL; Compound 31543 Calcitriol - 20 μg/mL; Compound 31543 Calcitriol - 40 μg/mL; Compound 31543 Calcitriol - 60 μg/mL; Compound 31543 Calcitriol - 80 μg/mL: BPM1543 Calcitriol, Topical application, 0.25 mL to be applied to each of the four quadrants of the scalp twice daily, morning and night with 10-14 hours between applications
Arm/Group | Compound 31543 Calcitriol - 5 μg/mL | Compound 31543 Calcitriol - 10 μg/mL | Compound 31543 Calcitriol - 20 μg/mL | Compound 31543 Calcitriol - 40 μg/mL | Compound 31543 Calcitriol - 60 μg/mL | Compound 31543 Calcitriol - 80 μg/mL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/6 | 4/4 | 1/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 4/4 | 3/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compound 31543 Calcitriol - 5 μg/mL (N=3) | Compound 31543 Calcitriol - 10 μg/mL (N=3) | Compound 31543 Calcitriol - 20 μg/mL (N=6) | Compound 31543 Calcitriol - 40 μg/mL (N=4) | Compound 31543 Calcitriol - 60 μg/mL (N=4) | Compound 31543 Calcitriol - 80 μg/mL (N=3)
Supraventicular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehyrdation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compound 31543 Calcitriol - 5 μg/mL (N=3) | Compound 31543 Calcitriol - 10 μg/mL (N=3) | Compound 31543 Calcitriol - 20 μg/mL (N=6) | Compound 31543 Calcitriol - 40 μg/mL (N=4) | Compound 31543 Calcitriol - 60 μg/mL (N=4) | Compound 31543 Calcitriol - 80 μg/mL (N=3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vitamin D Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The tables in this report reflect safety and effectiveness data to the best knowledge of the sponsor.

However, the results were generated from partially audited data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT01588522/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT01588522/SAP_001.pdf